CLINICAL TRIAL: NCT05398055
Title: Efficacy of Azithromycin Plus Doxycycline Compared to Doxycycline Plus Placebo in Patients With Rocky Mountain Spotted Fever in Hospital General de Mexicali of ISESALUD and Hospital General No. 30 Instituto Mexicano Del Seguro Social
Brief Title: Efficacy of Azithromycin Plus Doxycycline Versus Doxycycline Plus Placebo in Patients With Rocky Mountain Spotted Fever
Acronym: Rocky-Z
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexicali (Other)
Responsible Party: Principal Investigator, Hiram Jaramillo Ramirez, Clinical professor, Hospital General de Mexicali
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-01//2022-05-09-066-20
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Rocky Mountain Spotted Fever
Keywords: Rocky Mountain Spotted Fever; Azithromycin; Doxycycline
MeSH Terms: conditions — Rocky Mountain Spotted Fever | interventions — Azithromycin; Doxycycline

STUDY DESIGN:
Intervention Model Description: Controlled randomized trial with placebo, triple blinded, multicenter study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized through the program ¨Randomizer for Clinical Trial¨ to be assigned in group of treatment A or B. One of the treatments will be azithromycin 500 mg orally every 24 hours for three dose plus doxycycline 100 mg orally every 12 hours for 7 days and the other schedule it will be doxycycline 100 mg orally every 12 hours for 7 days plus placebo 1 capsule every 24 hours, 3 doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Azithromycine group
  Interventions: Drug: Azithromycin + Doxycycline
- B (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo + Doxycycline

INTERVENTIONS:
Drug: Azithromycin + Doxycycline — azithromycin 500 mg orally every 24 hours for three dose plus doxycycline 100 mg orally every 12 hours for 7 days
  Other Names: A
  Arms: A
Drug: Placebo + Doxycycline — doxycycline 100 mg orally every 12 hours for 7 days plus placebo 1 capsule every 24 hours, 3 doses
  Other Names: B
  Arms: B

SUMMARY:
The aim of this study is to impove the pharmacological treatment of Rocky mountain spotted fever, since is a very ancient disease with an antibiotic therapy that have not changed much the mortality rates, being compared with the natural curse of the disease.

DETAILED DESCRIPTION:
Rocky mountain spotted fever is a potentially fatal infectious disease wich is transmitted trough vectors. This particular infection is caused by Rickettsia rickettsii wich is a gramnegative intracellular bacilli. The pathophysiological mechanism and clinical manifestation is mainly due to the vascular affectation, since this pathogen has a tropism for endothelial cells. As it has been mentioned, this is an obligate intracellular pathogen, so the main choice with the antibiotic therapy is tetracyclines because of its action mechanism in the inhibition of the subunit 30S. The objective of the study is to prove new strategies of treatment to improve the pharmacological aproach by implementing Azithromycin, wich is a macrolide that inhibits de 50S subunit of the bacteria. Azithromycin has shown effectivity against other rickettsial diseases.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Over 18 years old
* hospitalized in the internal medicine service, emergency department or intensive care unit of Hospital General de Mexicali (ISESALUD) or Hospital General Zona No. 30 (IMSS) with suspicion of RMSF that present fever and 2 or more of the next symptoms: headache, myalgia, rash, nausea, pharyngeal hyperemia, vomiting, abdominal pain, neurological disorders.
* In addition to at least one of the next epidemiologycal fators: presence of vectors in areas of residence or endemic areas visited two weeks prior to the onset of symptoms, history of visiting or residing in areas with RMSF transmission in the last two weeks, existence of confirmed cases in the locality of origin, history of vector bite or contact with dogs in the two weeks.

Exclusion Criteria:

* Other clinical suspicion rather than RMSF
* History of allergy to doxycycline, azithromycin, bean starch or bovine gelatin.
* Not signing the informed consent
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality of azithromycin plus doxycycline vs doxycycline plus placebo | 3 years

SECONDARY OUTCOMES:
Number of hospitalization days in each arm | 3 years
Number of participants with renal replacement therapy. | 3 years
Number of participants that required amines in both groups. | 3 years
Number of fever days in both arms. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiram J Jaramillo-Ramirez, MD, Principal Investigator — Hospital General de Mexicali
Locations (1):
- Hospital General de Mexicali, Mexicali, Estado de Baja California, Mexico